CLINICAL TRIAL: NCT07243977
Title: Comparison of Efficacy of Microneedling Along With Topical Vitamin D3 Versus Microneedling Alone in the Treatment of Alopecia Areata
Brief Title: Comparison of Microneedling Along With Topical Vitamin D3 Versus Microneedling in Alopecia Areata
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Rameen Masood, Principal Investigator, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ServicesIMSP1
Record Dates: First submitted 2025-09-21; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-09

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata; Autoimmune Hair Loss; Microneedling; Hair Follicle Regeneration
MeSH Terms: conditions — Alopecia Areata | interventions — Percutaneous Collagen Induction; Cholecalciferol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Microneedling + Vitamin D3 (Experimental): Received microneedling with a dermapen (needle length 1.5-2 mm, highest speed level 4-5) performed until pinpoint bleeding appeared, combined with topical vitamin D3 application (Sunny D3® 200,000 IU/1 ml, aqueous preparation). Half the dose of vitamin D3 was applied before microneedling and the remaining after the procedure. Maximum dose used per session was 2.5 mg (0.5 ml). Sessions were repeated every 2 weeks for up to 6 sessions.
  Interventions: Procedure: Microneedling + Vitamin D3
- Group Microneedling Alone (Active Comparator): Received microneedling with a dermapen (needle length 1.5-2 mm, highest speed level 4-5) performed until pinpoint bleeding appeared, without vitamin D3 application. Sessions were repeated every 2 weeks for up to 6 sessions.
  Interventions: Procedure: Microneedling

INTERVENTIONS:
Procedure: Microneedling + Vitamin D3 — Dermapen treatment with adjustable needle length (1.5-2 mm), performed under local anaesthesia until pinpoint bleeding appeared. Aqueous vitamin D3 solution (Sunny D3® 200,000 IU/1 ml, 5 mg/ml) applied topically before and after microneedling.
  Other Names: Cholecalciferol topical solution; Microneedling
  Arms: Group Microneedling + Vitamin D3
Procedure: Microneedling — Dermapen treatment with adjustable needle length (1.5-2 mm), performed under local anaesthesia until pinpoint bleeding appeared.
  Arms: Group Microneedling Alone

SUMMARY:
Alopecia areata is a common condition that causes sudden, patchy hair loss on the scalp and other body sites. It is believed to occur when the body's immune system mistakenly attacks the hair follicles, leading to hair loss that can range from small patches to more widespread involvement. While many treatments have been tried, including steroids and newer medicines, none offer a guaranteed permanent cure.

Microneedling is a technique in which very fine needles are used to create small punctures in the skin. This stimulates natural healing, improves blood supply to hair roots, and activates stem cells that support new hair growth. It also allows medicines applied to the skin to penetrate more effectively. Previous studies have shown that combining microneedling with certain topical medicines improves results compared to microneedling alone.

Vitamin D is known to play an important role in the regulation of the immune system and in the health of hair follicles. Applying vitamin D directly to the scalp after microneedling may enhance its effects, as the microchannels created by the needles allow the medicine to reach the deeper layers of the skin.

This study will compare two treatment approaches for patients with localized alopecia areata (affecting less than half of the scalp). One group will receive microneedling alone, while the other group will receive microneedling combined with topical vitamin D3. The treatments will be given every two weeks for a total of six sessions. Patients will then be followed for three months to see whether they achieve complete regrowth of hair in the affected areas, as measured by a standard scoring system for alopecia areata (SALT score).

The study will enroll 80 adults aged 18-60 years who have alopecia areata and have not received any recent treatment. By comparing these two approaches, the study aims to find out whether adding topical vitamin D3 to microneedling improves treatment outcomes. If effective, this combination could provide patients with a safe, affordable, and non-invasive option for treating alopecia areata.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Alopecia Areata and have not received any treatment for last 4 weeks.
* Age range of 18-60 years
* Both male and female patients

Exclusion Criteria:

* Active infection or atrophy of scalp due to previous treatment
* Patients with alopecia universalis or totalis.
* Pregnant or lactating mothers.
* Systemic co-morbidities like diabetes, hypertension, chronic liver or kidney disease and immunosuppression
* Unwilling or uncooperative patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2025-03-29 (Actual); Primary Completion 2025-09-29 (Actual); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving complete hair regrowth (S0 on SALT score) | 3 months after initiation of treatment (following up to 6 treatment sessions given at 2-week intervals).
  The Severity of Alopecia Tool (SALT) score will be used to measure the extent of scalp hair loss. The scale ranges from S0 (no hair loss, complete regrowth) to S5 (100% hair loss). Treatment will be considered effective if participants achieve S0 (complete hair regrowth with no hair loss) at the end of the study period compared with baseline assessment. Clinical photographs and dermoscopic findings will also be used to validate outcomes.

SECONDARY OUTCOMES:
Dermoscopic improvement in alopecia areata lesions. | From baseline to 3 months after treatment initiation
  Assessment of dermoscopic features with documentation of new vellus hair growth as an indicator of follicular regeneration.

CONTACTS AND LOCATIONS:
Overall Officials: Rameen Masood, Principal Investigator — Services Institute of Medical Sciences, Pakistan
Locations (1):
- Services Institute of Medical Sciences, Lahore, Lahore, Punjab Province, Pakistan